CLINICAL TRIAL: NCT05903014
Title: Effectiveness of N-Acetylcysteine in Motivational Enhancement Therapy for Nicotine Addiction: Study on the Dopaminergic Pathways, Changes in Functional Connectivity of fMRI Bold, and Changes in Smoking Abstinence
Brief Title: Effectiveness of N-Acetylcysteine (NAC) in Motivational Enhancement Therapy for Nicotine Addiction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Tribowo Tuahta Ginting Sugihen, SpKJ(K), Head of Psychiatry Departement Persahabatan National Hospital, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-06-0672
Record Dates: First submitted 2023-05-09; First posted 2023-06-15 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Nicotine Dependence; Nicotine Addiction
Keywords: Nicotine Dependence; Nicotine Addiction; NAC
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Acetylcysteine; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 3600 mg NAC per day in 12 weeks
  Interventions: Drug: n-acetylcysteine; Behavioral: Motivational Enhancement Therapy
- Placebo (Placebo Comparator): Placebo
  Interventions: Behavioral: Motivational Enhancement Therapy

INTERVENTIONS:
Drug: n-acetylcysteine — we give 3600 mg n-acetylcysteine divided twice a day, for 12 weeks
  Arms: Experimental
Behavioral: Motivational Enhancement Therapy — Motivational enhancement therapy with individual and/or group session to maintain and increase subject's motivation to quit smoking

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of the combination of n-acetylcysteine and motivational enhancement therapy on laboratory improvement in the form of changes in blood nicotine, radiological changes in the form of nerve connectivity on post-therapy frontostriatal fMRI examination and clinical changes in the form of abstinence, withdrawal symptoms and cravings in adult smoker.

DETAILED DESCRIPTION:
The main question it aims to answer are:

Obtain the effectiveness of combination of n-acetylcysteine and motivational enhancement therapy compared to a combination of motivational enhancement therapy and placebo on nicotine withdrawal symptom scores on nicotine addiction.

Obtaining the effectiveness of the combination of n-acetylcysteine and motivational enhancement therapy compared to the combination of motivational enhancement therapy and placebo on craving symptom scores on nicotine addiction.

Obtain the effectiveness of giving a combination of n-acetylcysteine and motivational enhancement therapy compared to a combination of motivational enhancement therapy and placebo in the incidence of abstinence in nicotine addiction.

Obtain the effectiveness of combination n-acetylcysteine and motivational enhancement therapy compared to a combination of motivational enhancement therapy and placebo on blood nicotine levels in nicotine addiction.

Obtain the effectiveness of combination n-acetylcysteine and motivational enhancement therapy compared to a combination of motivational enhancement therapy and placebo on n-acetylaspartate levels in the brain in nicotine addiction.

Obtain the effectiveness of combination n-acetylcysteine and motivational enhancement therapy compared to a combination of motivational enhancement therapy and placebo on glutamate levels in the brain on nicotine addiction.

Obtain an overview of nerve connectivity in nicotine addiction patient through post-therapy frontostriatal fMRI examination.

Evaluate the side effects and severe side effects of NAC administration on nicotine addiction.

Participants will:

Get blood testing for nicotine in 1st, 6th and 12th weeks Fill the QSU-Brief, MTWS questionnaire every 2 weeks for 12 weeks Get motivational enhancement therapy every 2 weeks for 12 weeks Get fMRI in the 12th week Consume 3600 mg n-acetylcysteine for 12 consecutive weeks (for treatment group) and placebo (for control group) Researchers will compare the laboratory, clinical and radiology improvement in both groups

ELIGIBILITY:
Inclusion Criteria:

1. Male or female who are active smokers are at least 18 years old and decide to stop smoking
2. Using tobacco cigarettes whether filtered or not
3. Active smoker for at least 6 months
4. Smoke at least 10 cigarettes per day
5. Currently in the preparation or action stage at the stage of changes
6. Able to follow instructions and research procedures

Exclusion Criteria:

Have/ suspected to have a systemic medical disorder or psychiatric disorder requiring acute management Currently using electronic cigarettes Currently using oral glucocorticoids Have an acute gastrointestinal ulcer Pregnant or breastfeeding or planning to become pregnant within the next 6 months Currently consume n-acetylcysteine Have a history of allergic reactions with n-acetylcysteine or its components Get therapy to stop smoking such as bupropion, varenicline or nicotine replacement therapy (NRT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of Abstinence | week 2
  number of patient that have been quick smoking at a specific period of time
Rate of Abstinence | week 4
  number of patient that have been quick smoking at a specific period of time
Rate of Abstinence | week 6
  number of patient that have been quick smoking at a specific period of time
Rate of Abstinence | week 8
  number of patient that have been quick smoking at a specific period of time
Rate of Abstinence | week 10
  number of patient that have been quick smoking at a specific period of time
Rate of Abstinence | week 12
  number of patient that have been quick smoking at a specific period of time
Score of Craving Symptoms | week 2
  Score is assessed with Brief Questionnaire of Smoking Urges Questionnaire. Higher score means higher urgency to smoke. Scale: 10-70
Score of Craving Symptoms | week 4
  Score is assessed with Brief Questionnaire of Smoking Urges Questionnaire. Higher score means higher urgency to smoke. Scale: 10-70
Score of Craving Symptoms | week 6
  Score is assessed with Brief Questionnaire of Smoking Urges Questionnaire. Higher score means higher urgency to smoke. Scale: 10-70
Score of Craving Symptoms | week 8
  Score is assessed with Brief Questionnaire of Smoking Urges Questionnaire. Higher score means higher urgency to smoke. Scale: 10-70
Score of Craving Symptoms | week 10
  Score is assessed with Brief Questionnaire of Smoking Urges Questionnaire. Higher score means higher urgency to smoke. Scale: 10-70
Score of Craving Symptoms | week 12
  Score is assessed with Brief Questionnaire of Smoking Urges Questionnaire. Higher score means higher urgency to smoke. Scale: 10-70
Score of Withdrawal Symptoms | week 2
  Score is assessed with Minnesota Tobacco Withdrawal Scale Questionnaire. Scale: 0-32. Higher score means higger withdrawal symtomps
Score of Withdrawal Symptoms | week 4
  Score is assessed with Minnesota Tobacco Withdrawal Scale Questionnaire. Higher score means higger withdrawal symtomps Scale: 0-32
Score of Withdrawal Symptoms | week 6
  Score is assessed with Minnesota Tobacco Withdrawal Scale Questionnaire. Higher score means higger withdrawal symtomps Scale: 0-32
Score of Withdrawal Symptoms | week 8
  Score is assessed with Minnesota Tobacco Withdrawal Scale Questionnaire. Higher score means higger withdrawal symtomps Scale: 0-32
Score of Withdrawal Symptoms | week 10
  Score is assessed with Minnesota Tobacco Withdrawal Scale Questionnaire. Higher score means higger withdrawal symtomps Scale: 0-32
Score of Withdrawal Symptoms | week 12
  Score is assessed with Minnesota Tobacco Withdrawal Scale Questionnaire. Higher score means higger withdrawal symtomps Scale: 0-32
Level of blood nicotine | week 6
  Level of blood nicotine
Level of blood nicotine | week 12
  Level of blood nicotine
level of n-acetylaspartate in Magnetic Resonance Spectroscopy (MRS) study | week 12
  level of n-acetylaspartate in Magnetic Resonance Spectroscopy (MRS) study
level of glutamate in Magnetic Resonance Spectroscopy (MRS) study | week 12
  level of glutamate in Magnetic Resonance Spectroscopy (MRS) study

SECONDARY OUTCOMES:
Side Effect of n-acetylcysteine consumption | every 2 weeks for 12 weeks
  Side Effect of n-acetylcysteine consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mottillo S, Filion KB, Belisle P, Joseph L, Gervais A, O'Loughlin J, Paradis G, Pihl R, Pilote L, Rinfret S, Tremblay M, Eisenberg MJ. Behavioural interventions for smoking cessation: a meta-analysis of randomized controlled trials. Eur Heart J. 2009 Mar;30(6):718-30. doi: 10.1093/eurheartj/ehn552. Epub 2008 Dec 24. PMID 19109354
- [Background] Schmaal L, Berk L, Hulstijn KP, Cousijn J, Wiers RW, van den Brink W. Efficacy of N-acetylcysteine in the treatment of nicotine dependence: a double-blind placebo-controlled pilot study. Eur Addict Res. 2011;17(4):211-6. doi: 10.1159/000327682. Epub 2011 May 24. PMID 21606648
- [Background] Prado E, Maes M, Piccoli LG, Baracat M, Barbosa DS, Franco O, Dodd S, Berk M, Vargas Nunes SO. N-acetylcysteine for therapy-resistant tobacco use disorder: a pilot study. Redox Rep. 2015 Sep;20(5):215-22. doi: 10.1179/1351000215Y.0000000004. Epub 2015 Mar 2. PMID 25729878
- [Background] Schulte M, Goudriaan AE, Kaag AM, Kooi DP, van den Brink W, Wiers RW, Schmaal L. The effect of N-acetylcysteine on brain glutamate and gamma-aminobutyric acid concentrations and on smoking cessation: A randomized, double-blind, placebo-controlled trial. J Psychopharmacol. 2017 Oct;31(10):1377-1379. doi: 10.1177/0269881117730660. Epub 2017 Sep 19. PMID 28922968
- [Background] Machado RCBR, Vargas HO, Baracat MM, Urbano MR, Verri WA Jr, Porcu M, Nunes SOV. N-acetylcysteine as an adjunctive treatment for smoking cessation: a randomized clinical trial. Braz J Psychiatry. 2020 Sep-Oct;42(5):519-526. doi: 10.1590/1516-4446-2019-0753. PMID 32725102
- [Background] Froeliger B, McConnell PA, Stankeviciute N, McClure EA, Kalivas PW, Gray KM. The effects of N-Acetylcysteine on frontostriatal resting-state functional connectivity, withdrawal symptoms and smoking abstinence: A double-blind, placebo-controlled fMRI pilot study. Drug Alcohol Depend. 2015 Nov 1;156:234-242. doi: 10.1016/j.drugalcdep.2015.09.021. Epub 2015 Sep 26. PMID 26454838
- [Background] McClure EA, Baker NL, Gipson CD, Carpenter MJ, Roper AP, Froeliger BE, Kalivas PW, Gray KM. An open-label pilot trial of N-acetylcysteine and varenicline in adult cigarette smokers. Am J Drug Alcohol Abuse. 2015 Jan;41(1):52-6. doi: 10.3109/00952990.2014.933839. Epub 2014 Jul 25. PMID 25062287
- [Background] Bernardo M, Dodd S, Gama CS, Copolov DL, Dean O, Kohlmann K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Bush AI, Berk M. Effects of N-acetylcysteine on substance use in bipolar disorder: A randomised placebo-controlled clinical trial. Acta Neuropsychiatr. 2009 Dec;21(6):285-91. doi: 10.1111/j.1601-5215.2009.00397.x. PMID 25384734
- [Background] Knackstedt LA, LaRowe S, Mardikian P, Malcolm R, Upadhyaya H, Hedden S, Markou A, Kalivas PW. The role of cystine-glutamate exchange in nicotine dependence in rats and humans. Biol Psychiatry. 2009 May 15;65(10):841-5. doi: 10.1016/j.biopsych.2008.10.040. Epub 2008 Dec 21. PMID 19103434